CLINICAL TRIAL: NCT04389775
Title: A Phase 1, Randomised, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of XW003 Injection in Healthy Adult Participants
Brief Title: To Evaluate the Safety, Tolerability, PK, and PD of XW003 Injection in Healthy Adult Participants
Acronym: XW003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sciwind Biosciences APAC CO Pty. Ltd. (Industry)
Collaborators: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SCW0502-1011/1012; ACTRN12620000344998 (Registry Identifier: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2020-03-24; First posted 2020-05-15 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Nonalcoholic Steatohepatitis
Keywords: Type 2 Diabetes Mellitus; Obesity; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: One of up to six (6) sequential cohorts (Cohorts A1 to A6). Participants in each cohort will be randomised to receive a single subcutaneous (SC) dose of either XW003 or matching placebo on Day 1 following an overnight fast. Two sentinel participants will receive a single SC dose of XW003 initially. If dosing of these sentinel participants proceeds without clinically significant safety signals in the first 48 hours post-dose, the remaining participants will receive a single dose of XW003 or placebo according to the randomisation schedule.
  Participants in Cohorts B1 to B3 (n=10 per cohort) will be randomized to receive a single SC dose of either XW003 (n=8) or matching placebo (n=2) once weekly for 6 weeks. Doses will be administered following an overnight fast of at least 10 hours.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A (Experimental): Subcutaneously administer a single dose of XW003, ranging from 0.03mg to 1.0mg, every cohort by the body weight.
  Interventions: Drug: Cohort A
- Placebo A (Placebo Comparator): Subcutaneously administer a single dose of volume-matching placebo, ranging from 0.03mg to 1.0mg, every cohort by the body weight.
  Interventions: Drug: Placebo A
- Cohort B (Experimental): Subcutaneously administer multiple SC doses of XW003, ranging from 0.2mg to 0.6mg, once weekly for 6 weeks.
  Interventions: Drug: Cohort B
- Placebo B (Placebo Comparator): Subcutaneously administer multiple SC doses of volume-matching placebo, ranging from 0.2mg to 0.6mg, once weekly for 6 weeks.
  Interventions: Drug: Placebo B

INTERVENTIONS:
Drug: Cohort A — Participants in each cohort (A1 to A6) will be randomised to receive a SC dose of XW003 on Day 1 after overnight fasting by body weight range:
  1. Proposed XW003 Dose Levels (50 kg-75 kg): 0.03mg, 0.1mg, 0.2mg, 0.4mg, 0.8mg and 0.6mg respectively for Cohorts A1 to A6.
  2. Proposed XW003 Dose Levels (76 kg-90 kg): 0.03mg, 0.1mg, 0.25mg, 0.5mg, 1.0 mg and 0.6mg.
  These doses are subject to change following SRC review of each cohort - XW003 dose level will not exceed 2.0 mg.
  Other Names: GLP-1 analogue
  Arms: Cohort A
Drug: Placebo A — Participants in each cohort (A1 to A6) will be randomised to receive a SC dose of volume-matching placebo on Day 1 after overnight fasting by body weight range:
  1. Proposed Placebo Dose Levels (50 kg-75 kg): 0.03mg, 0.1mg, 0.2mg, 0.4mg, 0.8mg, and 0.6mg respectively for Cohorts A1 to A6.
  2. Proposed Placebo Dose Levels (76 kg-90 kg): 0.03mg, 0.1mg, 0.25mg, 0.5mg, 1.0 mg and 0.6mg.
  These doses are subject to change following SRC review of each cohort - dose level will not exceed 2.0 mg.
  Other Names: Placebo
  Arms: Placebo A
Drug: Cohort B — Participants in cohorts B1 to B3 (n=10 per cohort) will receive multiple SC doses of XW003 (n=8) once weekly for 6 weeks following an overnight fast of at least 10 hours.
  1. Subject to change following SRC review of each cohort.
  2. Following 4 weeks of once weekly dosing, the SRC will review the safety data (and PK data for Cohort B1 only) to determine the treatment for the following cohort and whether dosing can commence in parallel.
  3. At least 3 days prior to Cohort B3 Week 3 (i.e., 3 days prior to the third dose in Cohort B3), the SRC will review the safety and PK data for Cohorts B1 and B2 to determine whether Cohort 3 dosing for Weeks 3 to 6 may commence.
  Other Names: GLP-1 analogue
  Arms: Cohort B
Drug: Placebo B — Participants in cohorts B1 to B3 (n=10 per cohort) will receive multiple SC doses of matching placebo (n=2) once weekly for 6 weeks following an overnight fast of at least 10 hours.
  1. Subject to change following SRC review of each cohort.
  2. Following 4 weeks of once weekly dosing, the SRC will review the safety data (and PK data for Cohort B1 only) to determine the treatment for the following cohort and whether dosing can commence in parallel.
  3. At least 3 days prior to Cohort B3 Week 3 (i.e., 3 days prior to the third dose in Cohort B3), the SRC will review the safety and PK data for Cohorts B1 and B2 to determine whether Cohort 3 dosing for Weeks 3 to 6 may commence.
  Other Names: Placebo
  Arms: Placebo B

SUMMARY:
XW003 is an acylated human GLP-1 analogue and is being development for diabetes mellitus, obesity and nonalcoholic steatohepatitis (NASH) management. This is a first-in-human (FIH), single-centre, double blind, randomised, SAD and MAD study of XW003 conducted in healthy adult participants. The study is designed to evaluate the safety, tolerability, PK, and PD of XW003 in healthy adult participants.

DETAILED DESCRIPTION:
Participants will undergo a Screening period beginning up to 28 days prior to randomisation/dose administration. Participants will undergo pre-dose assessments, post-dose assessments, and will complete an EOS follow-up visit or early termination (ET) visit.

Up to 42 participants will be enrolled into one of up to six (6) sequential cohorts (Cohorts A1 to A6). Participants in each cohort will be randomised to receive a single subcutaneous (SC) dose of either XW003 or matching placebo on Day 1 following an overnight fast. Two sentinel participants will receive a single SC dose of XW003 initially. If dosing of these sentinel participants proceeds without clinically significant safety signals in the first 48 hours post-dose, the remaining participants will receive a single dose of XW003 or placebo according to the randomisation schedule.

Participants in Cohorts B1 to B3 (n=10 per cohort) will be randomized to receive a single SC dose of either XW003 (n=8) or matching placebo (n=2) once weekly for 6 weeks. Doses will be administered following an overnight fast of at least 10 hours.

ELIGIBILITY:
Single Dose Cohort-Inclusion Criteria:

1. Healthy male or female participants, aged 18 to 55 years (inclusive at the time of informed consent);
2. Participants must be in good general health, with no significant medical history, have no clinically significant abnormalities on physical examination at Screening and/or before administration of study drug;
3. Participants must have a BMI greater than or equal to 20.0 kg/m2 and less than or equal to 35.0 kg/m2 and weigh greater than or equal to 50 kg but less than or equal to 90 kg at Screening;
4. Stable body weight for at least three (3) months prior to Screening (i.e., <5% change);
5. Participants must have A1c below 6.4%, FPG: 3.9 ~ 6.1 mmol/L (both inclusive) or 70~110 mg/dL (both inclusive). All other clinical laboratory values must be within normal range as specified by the testing laboratory, unless deemed not clinically significant by the Investigator or delegate;
6. Non-smoker and/or casual smoker who uses no more than 10 cigarettes (or equivalent quantity of any other nicotine containing products e.g., cigars, chewing tobacco, snuff, etc.) per week. Participants must abstain from smoking 5 days prior to admission and throughout the confinement period, and test negative on Day -1 for urine cotinine test. Participants must also abstain from smoking 72 hours prior to each outpatient visit;
7. Participants must agree to abstain from alcohol intake from 48 hours prior to admission and during the confinement period;
8. Women of childbearing potential (WOCBP) must be non-pregnant and must use an acceptable, highly effective double contraception from Screening until study completion, including the follow up period.
9. Males must not donate sperm for at least 90 days after the last dose of study drug;
10. Participants must have the ability and willingness to attend the necessary visits to the CRU;
11. Participants must be willing and able to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Single Dose Cohort-Exclusion Criteria:

1. Prior or ongoing medical conditions, medical history, physical findings, or laboratory abnormality that, in the Investigator's (or delegate's) opinion, may require treatment or render the participant unlikely to fully complete the study, or any condition that presents undue risk from the IP or procedures or interfere with study assessments;
2. Confirmed diagnosis of diabetes mellitus type 1, type 2, or of any other forms at any time, and/or occurrence of documented or suspected hypoglycaemic episodes within 12 months prior to Screening;
3. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2;
4. History of acute or chronic pancreatitis;
5. Participants must be willing not to undertake any strenuous exercise, including but not limited to weightlifting (greater than 5 times per week) within 5 days prior to first study drug administration and for the duration of the study (including the follow-up period);
6. Participants must not start or having started participation in any medical (e.g., assisted by a clinical dietician or nutritionist) or non-medical (e.g., by a gym coach) diet and/or exercise programme within 3 months prior to Screening and for the duration of the study (including the follow-up period);
7. Use and/or planned use of any approved or unapproved weight-lowering medication(s) (including but not limited to orlistat, sibutramine, rimonabant, phentermine, or liraglutide) and/or medical device(s) within 3 months prior to Screening and for the duration of the study (including the follow-up period);
8. Previous history of any major gastrointestinal (including hepatobiliary and/or pancreatic) surgeries, including but not limited to sleeve, subtotal, or total gastrectomy, gastrojejunostomy, gastroduodenectomy, gastroduodenostomy, jejunectomy, ileectomy (proto)colectomy, hepatectomy, and pancreatectomy (except for appendectomy or cholecystectomy) and planned performance of one or more of the above mentioned for the duration of the study (including the follow-up period);
9. History of cerebral stroke (including but not limited to cerebral infarction/hemorrhage) within 12 months prior to Screening;
10. History of acute coronary syndrome (angina pectoris/myocardial infarction) and any other major cardiac conditions (including but not limited to myocarditis, cardiac insufficiency/failure, and any clinically significant arrythmia[s]) within 12 months prior to Screening;
11. Systolic blood pressure (BP) greater than 140 mmHg and/or less than 90 mmHg and/or diastolic BP greater than 90 mmHg and/or less than 40 mmHg and/or pulse rate greater 100 bpm and/or less than 40 bpm at Screening with one repeat allowed per by the Investigator or delegate at Screening and/or on Admission
12. Any clinically significant arrhythmia(s) at Screening ECG; specifically, the participant's corrected QT interval (QTcF) (Fridericia's correction) is greater than 450 ms at Screening and on Day -1. An out-of-range or abnormal ECG may be repeated during Screening. On admission, three ECGs should be recorded consecutively, and the Investigator must evaluate the triplicate ECG. If the participant's QTcF is greater than 450 ms on at least two ECGs, the participant must be excluded;
13. Any medically uncontrolled respiratory disease(s) and/or condition(s), including but not limited to severe current asthma, chronic obstructive pulmonary disease, and obstructive sleep apnoea syndrome;
14. Fever (body temperature greater than 38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening;
15. Clinically significant gastrointestinal disease(s), including but not limited to inflammatory bowel disease, irritable bowel syndrome, celiac disease, dyspepsia, apparent diabetic gastroparesis, and diabetic diarrhoea;
16. With alanine aminotransferase (ALT), aspartate aminotransferase (AST), and/or alkaline phosphatase (ALP) greater than 1.5 × upper limit of normal (ULN) at Screening. Repeat testing at Screening is acceptable for out of range values following approval by the Investigator or delegate;
17. With a confirmed creatinine clearance (CLcr) using the Cockcroft-Gault equation below 90 mL/min. Repeat testing at Screening is acceptable for out of range values following approval by the Investigator or delegate;
18. History of clinically significant endocrine condition(s), including but not limited to hyper/hypothyroidism and/or hyper/hypoadrenalism;
19. History of primary or recurrent malignancy, except for non-melanoma skin cancer excised more than 2 years prior to Screening and/or cervical intraepithelial neoplasia having been successfully cured more than 5 years prior to Screening;
20. With clinically significant haematologic abnormalities, including but not limited to haemoglobin above 180 g/L and/or below 110 g/L, white blood cell count (WBC) above 10.5×10^9/L and/or below 3.5×10^9/L, absolute neutrophil count above 7.0×10^9/L and/or below 2.0×10^9/L, and/or platelet count above 300×10^9/L and/or below 130×10^9/L. Repeat testing at Screening is acceptable for out of range values following approval by the Investigator or delegate;
21. With any other clinically significant laboratory abnormalities in clinical biochemistry, coagulation function, and/or urinalysis. Repeat testing at Screening is acceptable for out of range values following approval by the Investigator or delegate;
22. With positive test result(s) for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening;
23. History of life-threatening infection (e.g. meningitis) and/or any major infections requiring parental antimicrobials within 6 months prior to Screening;
24. Regular alcohol consumption (by self-declaration) defined as greater than 21 alcohol units per week (where 1 unit = 284-mL of beer, 25-mL of 40% spirit or a 125-mL glass of wine). Participant is unwilling to abstain from alcohol beginning 48 hours prior to admission to the CRU and during the confinement period;
25. With a history of substance abuse or dependency in the last 12 months, or a history of recreational intravenous drug use over the last 5 years (by self-declaration);with a positive toxicology screening panel (urine test including qualitative identification of barbiturates, tetrahydrocannabinol [THC], amphetamines, methamphetamines, methylenedioxy-methamphetamine [MDMA], phencyclidine, benzodiazepines, opiates and cocaine), or alcohol breath test;
26. History of severe allergic or anaphylactic reactions;
27. Known or suspected intolerance or hypersensitivity to the IP, close related compounds, or any of the stated ingredients;
28. Blood donation or significant blood loss (greater than or equal to 400 mL) within 60 days prior to the first study drug administration;
29. Plasma donation within 7 days prior to the first study drug administration;
30. Being pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study and for at least 3 months after the last dose of study drug;
31. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half lives of the product (whichever is the longest) or participation in more than four investigational drug studies within 1 year prior to Screening;
32. Previous treatment with glucagon-like peptide 1 (GLP-1) agonists within the last 3 months;
33. Use of any prescription drug(s) and medical device(s) (other than hormonal contraception:

    OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring, or an IUD) within 2 weeks prior to the first study drug dosing or use of any over the-counter (OTC) medication, herbal remedies, supplements or vitamins within 1 week prior to the first study drug dosing and during the course of the study without prior approval of the Investigator and MM. Use of simple analgesic(s) (e.g., paracetamol, a nonsteroidal anti-inflammatory drug [NSAID]) may be permitted at the discretion of the Investigator;
34. Present comedication with drugs known to interfere with glucose metabolism, such as systemic corticosteroids, non-selective beta-blockers, and monoamine oxidase inhibitors;
35. Presence of any underlying physical and/or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the subject will comply with the protocol or complete the study per protocol.

Repeat Dose Cohort - Inclusion Criteria

To be eligible for this study, participants must meet all of the following additional inclusion criteria:

1. Participants must have a Body Mass Index (BMI) ≥24.0 kg/m2 and ≤34.0 kg/m2 and a Body weight ≥70 kg;
2. Participants must be willing to test and document glucose at home using a glucometer;

Repeat Dose Cohort - Exclusion Criteria:

A participant who meets any of the following additional exclusion criteria must be excluded from the study:

1. Obesity induced by endocrine disorders (e.g., Cushing Syndrome);
2. Any clinical laboratory values deviating from or outside the laboratory reference range unless considered not to be clinically significant by the Investigator or delegate;
3. History of thyroid tumors of family history of thyroid tumors.
4. Hemoglobin, white cell count, neutrophil count, and platelet count must fall within the laboratory's normal ranges. Any other hematological parameters outside the normal range may be acceptable if clinically insignificant and at the Investigator's discretion. Repeat testing at Screening is acceptable following approval by the Investigator or delegate;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-03-29 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From administration of XW003 on Day 1 to the last follow-up visit
  Count of adverse events

SECONDARY OUTCOMES:
Maximum observed XW003 plasma concentration | 36 days
  Calculated based on XW003 measured in blood.
Time of the maximum observed XW003 plasma concentration | 36 days
  Calculated based on XW003 measured in blood.
Area under the XW003 plasma concentration-time curve | 36 days
  Calculated based on XW003 measured in blood.
Apparent terminal half-life of XW003 | 36 days
  Calculated based on XW003 measured in blood.
Apparent terminal elimination rate constant of XW003 | 36 days
  Calculated based on XW003 measured in blood.
Apparent total clearance of XW003 | 36 days
  Calculated based on XW003 measured in blood.
Apparent volume of distribution of XW003 | 36 days
  Calculated based on XW003 measured in blood.
Change from Baseline in body weight | Day 36 for Cohort A and Day 71 for Cohort B
  Percentage of body weight loss
Change from Baseline in fasting plasma glucose | Day 36 for Cohort A and Day 71 for Cohort B
  Percentage of fasting plasma glucose change
Change from Baseline in plasma insulin and pro-insulin | Day 36 for Cohort A and Day 71 for Cohort B
  Percentage of plasma insulin and pro-insulin change
Change from Baseline in plasma C-peptide | Day 36 for Cohort A and Day 71 for Cohort B
  Percentage of plasma C-peptide change
Change from Baseline in plasma glucagon | Day 36 for Cohort A and Day 71 for Cohort B
  Percentage of plasma glucagon change
Change from Baseline in plasma lipids (triglyceride, low-density lipoprotein [LDL], and high-density lipoprotein [HDL]) | Day 36 for Cohort A and Day 71 for Cohort B
  Percentage of plasma lipids (triglyceride, low-density lipoprotein [LDL], and high-density lipoprotein [HDL]) change
Incidence of anti-XW003 antibodies at end of study | Pre-dose of XW003 on Day 1, end of study visit on Day 36 for Cohort A and Day 71 for Cohort B
  Count of episodes
Area under the plasma concentration curve time zero to the last detectable time point before second dose | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
Area under the plasma concentration curve over a dosing interval after first dosing | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
Maximum plasma concentration after first dosing | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
Time to maximum plasma concentration after first dosing | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
Terminal phase elimination rate-constant after first dosing | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
Terminal phase elimination half-life after first dosing | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
Clearance after last dosing | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
Volume of distribution after last dosing | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
AUC accumulation ratio constant | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts
Trough plasma XW003 concentrations before next dosing (Day 1 to last dosing) | 71 days
  Calculated based on XW003 measured in blood in repeat dose cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Snyder, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo W, Xu Z, Zou H, Li F, Li Y, Feng J, Zhu Z, Zheng Q, Zhu R, Wang B, Li Y, Hao S, Qin H, Jones CL, Adegbite E, Telusca L, Fenaux M, Zhong W, Junaidi MK, Xu S, Pan H. Discovery of ecnoglutide - A novel, long-acting, cAMP-biased glucagon-like peptide-1 (GLP-1) analog. Mol Metab. 2023 Sep;75:101762. doi: 10.1016/j.molmet.2023.101762. Epub 2023 Jun 24. PMID 37364710